CLINICAL TRIAL: NCT05303103
Title: Using Mixed-methods Approach to Explore the Long-term Effects of COVID-19: Presentations, Associating Factors, and Survivor Experience
Brief Title: Using Mixed-methods Approach to Explore the Long-term Effects of COVID-19
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Min-Sheng General Hospital (Other); National Yang Ming Chiao Tung University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202106071RINB
Record Dates: First submitted 2021-12-02; First posted 2022-03-31 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-06

CONDITIONS: Covid19
Keywords: Severe acute respiratory syndrome-coronavirus; long-term effects; mixed-methods; health-related quality of life; longitudinal cohort study
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Researchers warned that up to 80% of the survivors may experience multiple and severe long-term symptoms, sometimes called Long Coronavirus Disease(Long COVID). These Long COVID can persist for longer than three months and cause profound distress and life interferences.

The specific aims are to (1) integrate the state of science of Long COVID, (2) describe the changes of various symptoms and HRQOL(Health-related Quality of Life) after 3, 6, 9, and 12 months of COVID-19 diagnosis, (3) explore predicting factors of the existence and severity of Long COVID, and (4) explore how patient experienced COVID-19 symptoms.

It is a mixed-methods research project with embedded design. Among the three research stages, a systematical review will be conducted first to address aim one. In stage two, a longitudinal cohort study will be carried out to recruit and follow up with individuals diagnosed with COVID-19 for a year. During the follow-up, the participants will need to report their symptoms via online questionnaire, phone or video interviews. Those who did experience COVID-19 symptoms will be invited to join stage three study. Stage three is a qualitative descriptive study addressing aim 4.

Participants and recruitment. For stage two, the inclusion criteria are individuals who (1) are at least 20 years-old and (2) were diagnosed with COVID-19 within six months. Individuals who have cognitive impairment or other issues that prevents them from doing self-ratings of symptoms will be excluded.

Expecting outcomes. It is expected that Long COVID will pose huge burden on survivors and their families. This project can provide a solid reference to foresee possible problems in this population and formulate strategies for early detection and management.

DETAILED DESCRIPTION:
Background. When the COVID-19 pandemic sustains for more than a year, a growing number of COVID-19 survivors have returned to their community. However, researchers warned that up to 80% of the survivors may experience multiple and severe long-term symptoms, sometimes called Long COVID, even the subjects were asymptomatic or only had mild symptoms at diagnosis. These Long COVID can persist for longer than three months and cause profound distress and life interferences. Findings from studies and patient reports on social media suggest that various symptoms may be experienced, including fatigue, neurological symptoms, respiratory symptoms, and cardiovascular symptoms. With that being said, more areas, such as how Long COVID evolved after diagnosis, how investigators identify risk groups, and what are these survivors' needs, remain unclear. Aim. The overarching goal of this research project is to investigate the presentations and associating factors regarding Long COVID, and to explore survivor experience. The specific aims are to (1) integrate the state of science of Long COVID, (2) describe the changes of various symptoms and HRQOL after 3, 6, 9, and 12 months of COVID-19 diagnosis, (3) explore predicting factors of the existence and severity of Long COVID, and (4) explore how patient experienced COVID-19 symptoms. Design. It is a mixed-methods research project with embedded design. Among the three research stages, a systematical review will be conducted first to address aim one. In stage two, a longitudinal cohort study will be carried out to recruit and follow up with individuals diagnosed with COVID-19 for a year. During the follow-up, the participants will need to report their symptoms via online questionnaire, phone or video interviews (aim 2 and 3). Those who did experience COVID-19 symptoms will be invited to join stage three study. Stage three is a qualitative descriptive study addressing aim 4. Participants and recruitment. For stage two, the inclusion criteria are individuals who (1) are at least 20 years-old and (2) were diagnosed with COVID-19 within six months. Individuals who have cognitive impairment or other issues that prevents them from doing self-ratings of symptoms will be excluded. Potential participants will be identified through recruitment messages posting on social media and referrals from collaborating healthcare providers. Expecting outcomes. It is expected that Long COVID will pose huge burden on survivors and their families. This project can provide a solid reference to foresee possible problems in this population and formulate strategies for early detection and management. It is one of the few, if there is any, longitudinal study following up with COVID-19 survivors and including patients' perspectives.

ELIGIBILITY:
Inclusion Criteria:

* at least 20 years-old
* diagnosed with COVID-19 within six months

Exclusion Criteria:

* are still in the active phase of COVID-19 infection (i.e., diagnosed within 4 weeks)
* have cognitive impairment or other issues that prevents them from doing self-ratings of symptoms via phone interviews

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Potential subjects will be identified through the following strategies: (1) searching the intranet of participating medical institutions (e.g., National Taiwan University Hospital, National Yang Ming Chiao Tung University Hospital and Min-Sheng General Hospital), (2) recruitment messages posting on social media, and (3) referrals from collaborating healthcare providers.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2021-11-18 (Actual); Primary Completion 2023-06-24 (Actual); Study Completion 2023-06-24 (Actual)

PRIMARY OUTCOMES:
By exploring the predicting factors, individuals with high-risk of developing severe Long COVID can be identified and targeted early. | After 3 months of COVID-19 diagnosis.
  The investigators propose to use the combination of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core model (Taiwan Chinese version) and Quality of Life Questionnaire-Lung Cancer model (Taiwan Chinese version) to measure Long COVID symptoms.
  It consists of 30 items and measures patients' functions and symptoms by 4-point Likert scales, it also measures quality-of-life by 7-point Likert scale. While the lung cancer model consists of 29 items, the sub-scales of 'fear of progression (2 items)' and 'surgery-related problems (5 items)' will not be used as they are related to cancer progression and treatment. A 4-point Likert scale will rate the remanding 22 items in this study to measure additional symptoms. Higher scores for symptom scales represent more intense symptoms while higher scores for function scales and quality of life mean better function and quality level.
By exploring the predicting factors, individuals with high-risk of developing severe Long COVID can be identified and targeted early. | After 6 months of COVID-19 diagnosis.
  The investigators propose to use the combination of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core model (Taiwan Chinese version) and Quality of Life Questionnaire-Lung Cancer model (Taiwan Chinese version) to measure Long COVID symptoms.
  It consists of 30 items and measures patients' functions and symptoms by 4-point Likert scales, it also measures quality-of-life by 7-point Likert scale. While the lung cancer model consists of 29 items, the sub-scales of 'fear of progression (2 items)' and 'surgery-related problems (5 items)' will not be used as they are related to cancer progression and treatment. A 4-point Likert scale will rate the remanding 22 items in this study to measure additional symptoms. Higher scores for symptom scales represent more intense symptoms while higher scores for function scales and quality of life mean better function and quality level.
By exploring the predicting factors, individuals with high-risk of developing severe Long COVID can be identified and targeted early. | After 9 months of COVID-19 diagnosis.
  The investigators propose to use the combination of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core model (Taiwan Chinese version) and Quality of Life Questionnaire-Lung Cancer model (Taiwan Chinese version) to measure Long COVID symptoms.
  It consists of 30 items and measures patients' functions and symptoms by 4-point Likert scales, it also measures quality-of-life by 7-point Likert scale. While the lung cancer model consists of 29 items, the sub-scales of 'fear of progression (2 items)' and 'surgery-related problems (5 items)' will not be used as they are related to cancer progression and treatment. A 4-point Likert scale will rate the remanding 22 items in this study to measure additional symptoms. Higher scores for symptom scales represent more intense symptoms while higher scores for function scales and quality of life mean better function and quality level.
By exploring the predicting factors, individuals with high-risk of developing severe Long COVID can be identified and targeted early. | After 12 months of COVID-19 diagnosis.
  The investigators propose to use the combination of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-core model (Taiwan Chinese version) and Quality of Life Questionnaire-Lung Cancer model (Taiwan Chinese version) to measure Long COVID symptoms.
  It consists of 30 items and measures patients' functions and symptoms by 4-point Likert scales, it also measures quality-of-life by 7-point Likert scale. While the lung cancer model consists of 29 items, the sub-scales of 'fear of progression (2 items)' and 'surgery-related problems (5 items)' will not be used as they are related to cancer progression and treatment. A 4-point Likert scale will rate the remanding 22 items in this study to measure additional symptoms. Higher scores for symptom scales represent more intense symptoms while higher scores for function scales and quality of life mean better function and quality level.

SECONDARY OUTCOMES:
Enhance our understanding toward patient experience and can be used to design more patient- or family-centered care. | After 3 months.
  Investigators want to provide a fundamental and straightforward description regarding the survivors' symptoms and experiences. The qualitative results based on patient perspectives may provide a reference for selecting appropriate strategies of observing and documenting Long COVID.

CONTACTS AND LOCATIONS:
Overall Officials: Chia Chun Tang, PhD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tang CC, Wu WW, Ho SJ, Liu WD, Pan MY, Chang SC, Wang WS, Yeh YC, Chen CH, Chang JC. Clinically Significant Functional Impairments and Symptoms in COVID-19 Survivors: Empirical Research Quantitative. J Clin Nurs. 2025 Nov;34(11):4664-4672. doi: 10.1111/jocn.17715. Epub 2025 Mar 14. PMID 40084807

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/03/NCT05303103/Prot_SAP_000.pdf